CLINICAL TRIAL: NCT04626687
Title: Paclitaxel Coated Coronary Balloon Catheter in Treatment of Coronary Small Vessel Diseases
Brief Title: ACOART Paclitaxel SVD:Paclitaxel Coated Coronary Balloon Catheter in Treatment of Coronary Small Vessel Diseases
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Acotec Scientific Co., Ltd (Industry)
Collaborators: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACOART paclitaxel SVD
Record Dates: First submitted 2020-11-04; First posted 2020-11-12 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-07

CONDITIONS: Coronary Disease
Keywords: coronary small vessel diseases; DCB
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test DCB group (Experimental): use the DCB made by Acotec Scientific
  Interventions: Device: test DCB
- RESTORE DCB group (Active Comparator): use the DCB made by CARDIONOVUM GmbH
  Interventions: Device: RESTORE DCB

INTERVENTIONS:
Device: test DCB — use paclitaxel coated coronary balloon catheters to treat SVD
  Arms: test DCB group
Device: RESTORE DCB — use paclitaxel coated coronary balloon catheters(RESTORE DCB) with NMPA approval indication for treating SVD
  Arms: RESTORE DCB group

SUMMARY:
The purpose of the trial is to determine whether DCB made by Acotec Scientific is not inferior to RESTORE DEB made by CARDIONOVUM GmbH in treatment of small vessel coronary disease.

DETAILED DESCRIPTION:
This is a prospective, multi-center, randomized-controlled clinical trial to verify the efficacy and safety of DCB made by Acotec Scientific versus RESTORE DEB in treatment of small vessel coronary disease. And the primary endpoint is angiographic restenosis at 9 months post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years of age
* Subjects with symptomatic coronary artery disease with stable and unstable angina pectoris or secondary evaluation of stenosis after acute myocardial infarction (MI) and asymptomatic subjects with coronary atherosclerotic stenosis causing myocardial ischemia determined by the investigator
* Subjects with single, de novo lesion with stenosis of more than 70% (or more than 50% combined with symptoms of ischemia) in a vessel with visually estimated reference vessel diameter (RVD) ≥ 2.00 mm and ≤ 2.75 mm, and ≤ 26 mm in length.
* Subject must agree to clinical follow-up at 1, 6, 9, 12 months, and angiographic follow-up at 9 months.
* Subject can understand the study objectives psychologically and linguistically and shows sufficient compliance to the study protocol. Subjects express acceptance of the risks and benefits described in the informed consent form.

Exclusion Criteria:

* AMI within 1 week.
* Subject has congestive heart failure or NYHA IV.
* Subject with LVEF < 35%.
* Subject has undergone heart transplantation.
* Subject has cardiac arrhythmias, such as high-risk ventricular premature beat and/or ventricular tachycardia.
* Subject suffered stroke, gastrointestinal bleeding or active ulcer within the past 6 months, or with conditions associated with high risk of bleeding.
* Subject with a history of leukopenia (white blood cell count of < 3×109/L for >3 days), neutropenia (ANC<1000/mm3 for >3 days) or thrombocytopenia (platelet <100,000/mm3).
* Known renal insufficiency (eGFR<30 ml/min).
* Subject who is forbidden to use anticoagulation agents or anti-platelet drugs, and tolerate Aspirin or Clopidogrel.
* Life expectancy less than 12 months, or subjects who cannot complete 12-month follow-up.
* Pregnant or nursing subjects and those who plan pregnancy in the period up to 1 year following index procedure.
* Subject is currently participating in another investigational drug or device study that has not yet completed its primary endpoint.
* Subject unsuitable for study according to the investigator due to the investigator due to other reasons related to diseases.
* Angiography exclusions:Target lesion: Total occlusion lesion (TIMI 0), heavy calcified lesion that cannot be successfully dilated, bifurcation lesion (side branch ≥ 2.0 mm in diameter), restenosis lesion, thrombotic lesion, or left main disease;Non-target lesion: More than 2 non-target lesions or non-target lesion cannot be successfully treated.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Estimated)
Dates: Start 2021-04-06 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Angiographic percent diameter stenosis | at 9 months post-procedure
  (1-Segmental minimum lumen diameter [MLD]/ segmental reference vessel diameter [RVD]) ×100%

SECONDARY OUTCOMES:
Acute success | in the procedure
  Including instrument success rate, lesion success rate and surgical success rate
Rate of target lesion failure | within 12 months post-procedure
  A composite of cardiac death, target-vessel related myocardial infarction, and ischemia-driven target lesion revascularization
Diameter stenosis in-device | at 9 months post-procedure
  (1-the minimum cavity diameter of the device [MLD] / the reference vessel diameter of the device [RVD]) ×100%
Late lumen loss | at 9 months post-procedure
  Loss of late lumen in the segment and device

CONTACTS AND LOCATIONS:
Overall Officials: Xuebo Liu, MD, Principal Investigator — Shanghai Tongji Hospital, Tongji University School of Medicine
Locations (1):
- Shanghai Tongji Hospital, Tongji University School of Medicine, Shanghai, China